CLINICAL TRIAL: NCT03882645
Title: Diet, Exercise and Cardiovascular Health - Effects of Chinese Heart Healthy Diet on Blood Pressure Among People With High Cardiovascular Risk: a Parallel, Multicenter, Single-blind, Randomized Controlled Feeding Trial
Brief Title: Chinese Heart Healthy Diet for People With High Cardiovascular Risk in China (DECIDE-Diet)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment of the study participants
Sponsor: Peking University (Other)
Collaborators: Sun Yat-sen University (Other); Sichuan University (Other); Huadong Hospital (Other); Yangzhou University (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Yanfang Wang, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016YFC1300201
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Disease; Diet Modification; Randomized Controlled Trial
Keywords: Chinese Heart Healthy Diet; Randomized Controlled Trial; Feeding Study; Blood Pressure; serum lipids; Fasting Blood Glucose; Diet Modification
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, single-blind, parallel controlled intervention is proposed in this study. 360 subjects are anticipated to be enrolled from each research centers (Qingdao and Beijing, Shanghai, Guangzhou, Chengdu). After the one-week run-in period baseline information of eligible participants will be collected. Then the subjects will be allocated to intervention group or control group through central randomization. Subjects in intervention group will be given free CHH-Diet for four weeks, while the subjects in the control group will be given free usual diet conforming to local characteristics for four week.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of dietary intervention, it is impractical to blind the cook, dietitian and the study staff who are responsible for preparing the foods and taking all measurements of the diets. However, staffs conducting the outcome assessments will be blinded to the allocation of intervention assignments. In addition, every effort is made to blind the study participants to their intervention assignment. First, they will not be told of their group assignment. Second, the two groups will consume their meals in separate rooms. Third, the same dishes using similar food materials will be used for both groups at the same meal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHH-diet arm (Experimental): During the 4-week intervention period, free meals conformed to CHH-diet will be provided 3 times per daily (breakfast, lunch, dinner). Different center offers different meals of different cuisines but all conformed to "CHH-diet". The main nutrientional "healthy" goal of different cuisines will be achieved through specific nutrient targets, including fat, carbohydrate, protein, dietary fiber, sodium, potassium, magnesium and calcium.
  Interventions: Other: CHH-diet
- local usual diet arm (Other): During the 4-week intervention period, three meals per day (breakfast, lunch, dinner) will be provided free of charge in line with local dietary characteristics. The energy,protein, carbohydrate, as week as dietary fiber, sodium, calcium, magnesium and potassium will be kept the same as that in the run-in phase.
  Interventions: Other: local usual diet

INTERVENTIONS:
Other: CHH-diet — This study took the DASH Diet as the basic model and developed the "Chinese Heart Healthy Diet ( CHH-diet)" according to the principles in the "2016 Dietary Guidelines for Chinese Residents". The nutrients targets in CHH-diet are set as following: fat % of total kcal: 25-27% (saturated: 6%; monounsaturated: 12%; polyunsaturated: 8%); carbohydrate % of total kcal: 55-60%; protein % of total kcal: 17-19%; dietary fiber: 30 g/day; sodium: 3000 mg/day; potassium: 3700 mg/day; magnesium: 500 mg/day; calcium: 1200 mg/day. The total energy will be set according to how much participants are eating in run-in period.
  Arms: CHH-diet arm
Other: local usual diet — The nutrients targets and total energy in usual diet are set according to how much participants are eating in run-in period.
  Arms: local usual diet arm

SUMMARY:
The DECIDE - Diet (Diet, ExerCIse and carDiovascular hEalth - Chinese Heart Healthy Diet for People With High Cardiovascular Risk in China) is to evaluate the effects of CHH-diet in reducing blood pressure in Chinese people with high cardiovascular risk. The study will recruit 360 adults people from 4 centers in China. All eligible participants will participate in a 1-week run-in phase in which they are fed the usual Chinese diet. Participants who pass the run-in phase will be randomly assigned 1:1 to receive CHH-diet or usual diet with the use of a central concealed randomization procedure (simple randomization), stratified by center and batch.

The intervention will last 28 days. Primary outcome will be the change in systolic blood pressure. The secondary outcomes include the differences between the two groups in the changes of diastolic blood pressure, total cholesterol, fasting blood glucose, 10-year CVD risk, gut microbial community and food preference score.

DETAILED DESCRIPTION:
The Chinese Heart Healthy Diet (CHH-diet) is a study in the DECIDE project (Diet, ExerCIse and carDiovascular hEalth), which includes five studies. The others are DECIDE - Exercise, DECIDE - Salt in Elderly, DECIDE - Obesity in Children, and DECIDE - Smart Living. The primary aim of this study is to evaluate the effects of CHH-diet in reducing blood pressure in Chinese adults with high cardiovascular risk. The corresponding null hypothesis is the mean systolic blood pressure of participants in CHH-diet group is equal to the mean systolic blood pressure of those in usual diet group. The secondary aims of this study are: 1) to evaluate the effect of CHH-diet on reducing the blood lipid, blood glucose and overall risk of cardiovascular and cerebrovascular diseases; 2) the influence of different cuisines on the intervention effect; 3) the influence of baseline blood pressure, blood glucose and lipid levels on the intervention effect; 4) the difference of the food preference between the two groups; 5) the effect of CHH-diet on intestinal flora, and the influence of intestinal flora on the effect of CHH-diet on blood pressure, fasting blood glucose and blood lipids.

Potential participants will be evaluated for eligibility at each center located in cities accordance with the four cuisines: Qingdao and Beijing (Shandong cuisine), Shanghai (Huaiyang cuisine), Guangzhou (Cantonese cuisine), and Chengdu (Szechuan cuisine). Two screening visits will be performed to identify eligible participants. At the first visit, participants will be asked several key questions about inclusion and exclusion criteria. At the second visit, a full questionnaire and measurement will be conducted to screen eligible participants. All eligible participants will participate in a 1-week run-in phase in which they will be fed with the usual diet in urban China. A participant will be excluded if failing to consume more than three meals for any reason. Participants who pass the run-in phase will be re-check the inclusion and exclusion criteria and then assigned 1:1 to receive CHH-diet or usual diet with the use of a central concealed randomization procedure (simple randomization), stratified by center and batch after the each baseline survey completed. At each center, participants will enter the randomization phase through 3-4 batches according to the feeding capacity of each center.

Four different recipes of CHH-diet have been developed according to four local cuisines: Shandong cuisine (Qingdao and Beijing), Huaiyang cuisine (Shanghai), Cantonese cuisine (Guangzhou), and Chengdu (Szechuan cuisine), but the four different healthy recipes share the same nutrients targets. The control group will receive local usual diet with the similar 4-week menus as CHH-diet group, but their nutrients targets will be the same as run-in period. We will measure the actual intake of every meal for all participants during the whole study period to better estimate their nutrients intakes. All subjects will be advised to avoid outside food during the study period, and the information outside food should be reported if they eat.

Intake of foods and nutrients measurement: First, for each food/dish, raw food materials will be weighted after cleaning and before cooking. Then before the food served to the study participants it will also be weighted and recorded. After each meal, the leftover food from each participant will be measured and recorded as well. The average daily energy and dietary nutrient intake by each participants will be calculated using the China Food Composition (2nd Edition, volume 1).

The baseline data collection should be performed on the last two days of the run-in phase, which includes a questionnaire interview on demography, lifestyle and health behaviors, history of diseases, medication use (antihypertensive drugs, antidiabetic drugs, and lipid-lowering drugs), food preference; physical examinations (blood pressure, body weight & height, pulse rate); fasting blood tests (fasting glucose [FBG], total cholesterol [TC], low-density lipoprotein cholesterol [LDL-C], high-density lipoprotein cholesterol [HDL-C], triglycerides, and serum potassium); spot urine tests (sodium, potassium, creatinine excretion); and fecal sample tests on gut microbial community. The same physical examinations, medication use, food preference, fasting blood tests, spot urine tests, physical examinations and fecal sample tests on microbiome will be repeated at the end of the trial with the same methods by staffs blinded to the intervention. In addition, blood pressure, body weight, medication use, food preference assessment will be assessed weekly during the trial.

Power analysis: According to the findings from the DASH diet that successfully reduced SBP by 5.5 mmHg in 8 weeks, we conservatively assumed that CHH diet will reduce SBP by 3.0 mm Hg in comparison with the control diet in 4 weeks. And we further assumed the standard deviation of SBP change will be 8 mmHg in the control group according to our previous studies. To have 90% power with a type I error rate of 5% to detect the assumed effect size, we would need 165 participants in each arm. Assuming that 10% of study participants will be lost by the end of the study, we will recruit a total of 360 participants (90 from each center).

Statistical analysis: The primary analyses will follow the intention-to-treat principle and will be conducted among participants who have been randomized and the primary outcome are collected. The linear regression will be used to estimate the absolute differences between two groups in both primary and secondary outcomes, reported as least squared means after adjusting for centers. The differences in pre-set confounders between groups will be calculated by using a t-test, Wilcoxon rank test, or chi-square test. Sensitivity analyses will be performed to adjust for the imbalanced pre-set confounders if existed and to repeat the analyses with imputed missing values due to the lost to follow ups if the missing rates of outcomes higher than 5%. Per-protocol analyses will be conducted among population including those who consume more than 80% of study meals and completed the final follow up, with body weight change within 2kg and as well as the medications and dosages unchanged throughout study period. Subgroup analyses will be performed to identify potential modifiers of the intervention effect, including type of Chinese cuisine (center), gender, age, baseline multi-morbidity, medications use, blood pressure, glucose, total cholesterol, and estimated 10-year risk of ischemic cardiovascular disease.

Date management: a Web-based Data Management System (Redcap) will be used to facilitate data collection and central management during the whole process of the trial. Access to stored information is restricted to authorized personnel only. Paper forms with participant-identifiable information are held in secure, locked in file cabinets within a restricted area of each site.

Quality control: quality control team was established before the initiation of this study. All the researchers participating in this study must attend the technical training and pass the examination organized by the coordinating center, including study protocol, informed consent, case report form, standard operating procedures of participants' data collections, collection and preservation methods of biological samples. All biological samples will be tested in our central laboratory located in Beijing. The biochemist who performs the assessment will be blinded to allocation. In addition, 10% of urine and blood samples will be taken as split samples to control the quality of laboratory test results. On-site and on-line monitoring for data verification will be used. Each site will have at least two on-site monitoring visits, one at the beginning of the trial and one at the end of the trial. Quality control team will convene executive committee teleconferencing for quality control if necessary.

Data sharing plan: Data are available upon reasonable request (Yanfang Wang, pucri_wangyf1225@bjmu.edu.cn).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 25 and 75 years old.
2. Systolic blood pressure (SBP) in 130-159 mm Hg, regardless of medication use;
3. Living in this community for the past six months and without intention to move out or go out in the next three months.
4. Agree to keep the current drugs and their dosages unchanged throughout the study.
5. Promised to follow the study diets for 5 weeks, and eat at least 18 study meals per week.
6. Able to eat at least one meal per day at local research center.
7. Signed Informed consent.

Exclusion Criteria:

1. Fasting blood glucose ≥10.0 mmol/L.
2. Total cholesterol ≥7.2 mmol/L.
3. Any changes in dose and/or type of oral medication for antihypertensive, hypoglycemic or lipid-lowering in the past 3 months.
4. Insulin injection within 1 month.
5. Unable or unwilling to change diet for any reason (such as vegetarians).
6. Relatives of researchers or administrators.
7. Family members already in this study.
8. Alcohol consumption ≥ 8 drinks per week for women, ≥15 drinks per week for men.
9. BMI ≥ 30Kg/m2, or currently losing weight.
10. Acute cardiovascular and cerebrovascular events within the past 6 months.
11. A history of chronic kidney disease, intestinal irritation or asthma.
12. Current or planned pregnancy prior to end of study, or breast-feeding.
13. Other serious chronic disease thought to interfere with the effect of the diet or with participation, such as tumor, chronic heart failure, severe depression or other mental disorders, immobilization or unable to move freely.
14. Allergy of common food (e.g. eggs, seafood, peanuts, etc.).
15. On special diet due to medical needs.
16. Acute diseases such as upper respiratory tract infection, fever, severe diarrhea.
17. Deafness, dementia, and inability to communicate.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
The change on systolic blood pressure among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of systolic blood pressure in CHH-diet group compared with changes of usual diet group. Blood pressure will be taken 3 times within 24 hours at baseline and at the end of this trial: one in the morning between 8:00 am to 10:00 am, one in the afternoon between 2:00 pm to 4:00 pm, and one in the evening between 6:00 pm to 8:00 pm, respectively. In each time, 3 readings should be taken with at least one minute intervals. The mean of nine SBP readings will be used for the calculation of the changes in each participant.

SECONDARY OUTCOMES:
The change on the diastolic blood pressure among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the diastolic blood pressure in CHH-diet group compared with changes of usual diet group. Blood pressure will be taken 3 times within 24 hours at baseline and at the end of this trial: one in the morning between 8:00 am to 10:00 am, one in the afternoon between 2:00 pm to 4:00 pm, and one in the evening between 6:00 pm to 8:00 pm, respectively. In each time, 3 readings should be taken with at least one minute intervals. The mean of nine DBP readings will be used for the calculation of the changes in each participant.
The change on the serum total cholesterol among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the serum total cholesterol in CHH-diet group compared with changes of usual diet group. Blood sample of participants from the each center will be collected in their fasting state by qualified nurses. Centrifuged serum samples will be frozen and transported to Beijing through complete cold chain and measured in the central laboratory, Lawke Health Laboratory in Beijing.
The change on the fasting blood glucose among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the fasting blood glucose in CHH-diet group compared with changes of usual diet group. Blood sample of participants from each center will be collected in their fasting state by qualified nurses. Centrifuged serum samples will be frozen and transported to Beijing through complete cold chain and measured in the central laboratory, Lawke Health Laboratory in Beijing. Fasting blood glucose (using hexokinase method) will be carried out on a Roche Cobas c501 automatic biochemistry analyzer.
The change on 10-year CVD risk among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the 10-year CVD risk in CHH-diet group compared with changes of usual diet group. The 10-year CVD risk will be calculated according to 10-year risk prediction models for ischemic cardiovascular disease derived from the USA-PRC Collaborative Study of Cardiovascular Epidemiology cohort.
The change on food preference scores among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the food preference scores in CHH-diet group compared with changes of usual diet group. A visual analogue scale ranged from 0 to 10 was developed to assess the food preference.
The change on gut microbial community among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Faecal DNA will be extracted from each sample using the QIAamp Fast DNA Stool Mini Kit (QIAGEN, cat. 51604). To investigate the microbial community, shotgun metagenomic and amplicon sequencing strategies will be used.

OTHER OUTCOMES:
Dietary patterns analysis | up to 5 weeks (1 week run-in and 4 weeks intervention)
  The dietary patterns of the subjects in both groups were analyzed based on their individual intake of various foods during the study period.
The change on the serum LDL-C among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the serum LDL-C in CHH-diet group compared with changes of usual diet group.
  This outcome was moved from secondary outcome to other outcome because there are four outcomes of serum lipids profile and they are co-related to each other. We chose to keep one of them to reflect the change in serum lipids to reduce the type I error. In our previous experiences, total cholesterol is most reliably measured in labs among four lipid outcomes and more commonly used in clinical practice, partically in primary care. Thus we kept total cholesterol in secondary outcomes and moved other three lipid outcomes into other outcomes. The change was specified in the published protocol (BMJ Open 2020;10:e036394. doi:10.1136/bmjopen-2019-036394) without giving the reason described above in time.
The change on the serum HDL-C among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the serum HDL-C in CHH-diet group compared with changes of usual diet group.
  This outcome was moved from secondary outcome to other outcome because there are four outcomes of serum lipids profile and they are co-related to each other. We chose to keep one of them to reflect the change in serum lipids to reduce the type I error. In our previous experiences, total cholesterol is most reliably measured in labs among four lipid outcomes and more commonly used in clinical practice, partically in primary care. Thus we kept total cholesterol in secondary outcomes and moved other three lipid outcomes into other outcomes. The change was specified in the published protocol (BMJ Open 2020;10:e036394. doi:10.1136/bmjopen-2019-036394) without giving the reason described above in time.
The change on the serum TG among people at high risk of cardiovascular and cerebrovascular diseases | before and after 4-week intervention
  Changes of the serum TG in CHH-diet group compared with changes of usual diet group.
  This outcome was moved from secondary outcome to other outcome because there are four outcomes of serum lipids profile and they are co-related to each other. We chose to keep one of them to reflect the change in serum lipids to reduce the type I error. In our previous experiences, total cholesterol is most reliably measured in labs among four lipid outcomes and more commonly used in clinical practice, partically in primary care. Thus we kept total cholesterol in secondary outcomes and moved other three lipid outcomes into other outcomes. The change was specified in the published protocol (BMJ Open 2020;10:e036394. doi:10.1136/bmjopen-2019-036394) without giving the reason described above in time.

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Wang, Principal Investigator — Peking University
Locations (6):
- China (6):
  - Peking University, Beijing, Beijing Municipality
  - Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Clinical Research Institute, Qingdao, Shandong
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - Sichuan University, Chengdu, Sichuan
  - Peking Univeristy Clinical Research Institute, Beijing, string:China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie W, Wang Y, Sun J, Zeng G, Zhu H, Yang Z, Gao P, Yang J, Feng L, Lin PH, Li M, Xu J, Chen J, Wu Y. Protocol of a multicenter, single-blind, randomised, parallel controlled feeding trial evaluating the effect of a Chinese Healthy Heart (CHH) diet in lowering blood pressure and other cardiovascular risk factors. BMJ Open. 2020 Aug 20;10(8):e036394. doi: 10.1136/bmjopen-2019-036394. PMID 32819944
- [Background] Wang Y, Feng L, Zeng G, Zhu H, Sun J, Gao P, Yuan J, Lan X, Li S, Zhao Y, Chen X, Dong H, Chen S, Li Z, Zhu Y, Li M, Li X, Yang Z, Li H, Fang H, Xie G, Lin PH, Chen J, Wu Y; DECIDE-Diet Study Group. Effects of Cuisine-Based Chinese Heart-Healthy Diet in Lowering Blood Pressure Among Adults in China: Multicenter, Single-Blind, Randomized, Parallel Controlled Feeding Trial. Circulation. 2022 Jul 26;146(4):303-315. doi: 10.1161/CIRCULATIONAHA.122.059045. Epub 2022 Jul 11. PMID 35861850
- [Derived] Li Q, Feng L, Sun J, Zhu H, Zeng G, Gao P, Yuan J, Zhao Y, Li S, Lan X, Chen X, Li Z, Chen S, Dong H, Li M, Li X, Yang Z, Li H, Xie G, Wang Z, Lin PH, Chen J, Wang Y, Wu Y; DECIDE-Diet Study Group includes the following; Study Management Committee; Study Advisory Committee; Participating centers and staff information. Effects of Chinese heart-healthy diet on blood lipids, glucose, and estimated 10-y cardiovascular disease risk among Chinese adults: results on secondary outcomes of a randomized controlled trial. Am J Clin Nutr. 2024 Feb;119(2):333-343. doi: 10.1016/j.ajcnut.2023.12.008. Epub 2023 Dec 16. PMID 38110039